CLINICAL TRIAL: NCT01480661
Title: Analysis of Airway Responses in Severe COPD Patients to Daxas®, Using CT Based Functional Respiratory Imaging
Brief Title: Evaluation With CT Scan of Possible Changes in Airways After Treatment With Daxas® in Severe Chronic Obstructive Pulmonary Disease Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: FLUIDDA nv (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: FLUI-2011-77; 2011-004271-36 (EudraCT Number)
Record Dates: First submitted 2011-11-21; First posted 2011-11-29 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Computed Tomography scan; Functional Respiratory Imaging; Roflumilast; Health Related Quality of Life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roflumilast (Active Comparator)
  Interventions: Drug: Roflumilast; Radiation: Functional Respiratory Imaging
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo of Roflumilast; Radiation: Functional Respiratory Imaging

INTERVENTIONS:
Drug: Roflumilast — Roflumilast 500 µg, once a day in the morning during 6 months
  Other Names: Daxas®
  Arms: Roflumilast
Drug: Placebo of Roflumilast — Placebo 500 µg, once a day in the morning during 6 months
  Arms: Placebo
Radiation: Functional Respiratory Imaging — CT scan of thorax, at baseline and after 6 months

SUMMARY:
In this study the possible changes in airway geometry and function induced by 6 month oral treatment with Daxas® (roflumilast) will be evaluated. The use of functional respiratory imaging (FRI) on the phenotyping of chronic obstructive pulmonary disease (COPD) patients will be examined. The study population consists of 40 severe COPD patients, global initiative for chronic obstructive lung disease (GOLD) stages III until IV.

Imaging parameters will be assessed and the correlation with lung function and health related quality of life will be checked before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient ≥ 30 years old
* Patient with BMI ≥ 20
* Written informed consent obtained
* Female patient of childbearing potential who confirm that a contraception method was used at least 14 days before visit 1 and will continue to use a contraception method during the study.
* Patient should be treated according to GOLD guidelines
* COPD patient with GOLD stages III until IV
* Patient with smoking history of at least 10 pack-years
* Patient takes Spiriva® and a fixed combination of inhaled steroids and long acting beta agonist (LABA) at least 6 weeks before visit 1
* Patient must be able to understand and complete the protocol requirements, instructions, questionnaires and protocol-stated restrictions.

Exclusion Criteria:

* Pregnant or lactating females
* Patient with severe immunological diseases and/ or severe acute infectious diseases.
* Patient with heart failure
* Patient with diagnosis of cancer (except basal cell carcinoma)
* Patient with a history of depression associated with suicidal ideation or behaviour
* Patient with moderate or severe hepatic impairment.
* Patient with lactose intolerance
* Patient is unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study.
* Patient who received any investigational new drug within the last 4 weeks prior to the screening visit or twice the duration of the biological effect of any drug (whichever is longer).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Changes in airway geometry and function using CT based functional respiratory imaging. | At baseline and after 6 months of treatment
  The primary objective of this study is to evaluate the possible use of CT based functional respiratory imaging (CT-FRI) on the phenotyping of severe COPD patients after a 6 month treatment with Daxas®.

SECONDARY OUTCOMES:
Lung function tests (spirometry, bodyplethysmography, diffusion capacity, forced oscillation technique) | At baseline and after 6 months of treatment
  Imaging parameters will be assessed and the correlation with lung function will be checked before and after treatment.
Health related quality of life | At baseline and after 6 months of treatment
  Imaging parameters will be assessed and the correlation with health related quality of life will be checked before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Backer, MD, PhD, Principal Investigator — University Hospital, Antwerp; Lieven Bedert, MD, Principal Investigator — ZNA Middelheim
Locations (2):
- Belgium (2):
  - ZNA Middelheim, Antwerp, Antwerp
  - Antwerp University Hospital, Edegem, Antwerp